CLINICAL TRIAL: NCT00903669
Title: Anthropometric Angular Measurement to Determine Muscle Tonus in Patients With Peripheral Facial Paralysis
Acronym: PF
Status: Completed | Type: Observational
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Jorge Rizzato Paschoal, Department of Otolaryngology School of Medical Sciences - UNICAMP
Other Study IDs: ATessitore
Record Dates: First submitted 2009-05-14; First posted 2009-05-18 (Estimated); Last update posted 2009-05-18 (Estimated); Status verified 2009-05

CONDITIONS: Peripheral Facial Paralysis
Keywords: Facial paralysis; Muscle tonus; Rehabilitation; Myofunctional; Stomatognathic system
MeSH Terms: conditions — Facial Paralysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Peripheral Facial Paralysis (PFP): Patients who are diagnosed with peripheral facial paralysis.

SUMMARY:
The current study sought to determine the reliability of the rehabilitation protocol using the labial commissure angle (LCA) as an indicator of both muscle tonus and therapeutic success. The investigators hypothesized that this measurement would provide objective data regarding the efficacy of rehabilitation for these challenging patients.

DETAILED DESCRIPTION:
CONTEXT AND OBJECTIVE: In cases of peripheral facial paralysis (PFP), diminished facial movements and their resultant cosmetic sequelae may have significant emotional repercussions, in addition to producing pronounced functional deficits. Abnormal muscle proprioception and deviation of the nasal-labial filter may also interfere with articulation of the labiodental and bilabial phonemes, thus diminishing speech intelligibility. In relation to stomatognathic functions, weakened labial occlusion decreases intraoral pressure, thereby hindering liquid retention in the buccal cavity and giving rise to vestibular stasis on the paralyzed side. The aim of this study was to evaluate the reliability of the labial commissure angle (LCA) as an anthropometric marker for objectively assessing changes in facial muscle tonus.

ELIGIBILITY:
Inclusion Criteria:

* age range between 20 and 70 years
* incomplete PFP (Degree IV)
* integral facial nerve (FN)

Exclusion Criteria:

* systemic disease
* potentially aggravating the PFP (neurological, degenerative, endocrinological)

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with PFP treated in the Hospital of Unicamp
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2005-01; Primary Completion 2005-09 (Actual); Study Completion 2006-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge R Paschoal, Principal Investigator — Universidade Estadual de Campinas, Unicamp
Locations (1):
- Universidade estadual de Campinas, Campinas, São Paulo, Brazil